CLINICAL TRIAL: NCT05445986
Title: Clinical, Radiographic and Aesthetic Evaluation of Immediate Implant Placement With or Without Buccal Bone Dehiscence in the Anterior Maxilla
Brief Title: Immediate Implant Placement With or Without Buccal Bone Dehiscence
Status: Completed | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Junyu Shi, Principal Investigator, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: SH9H2022-136
Record Dates: First submitted 2022-06-27; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Dental Implant Failed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group1: socket with intact buccal bone plate
  Interventions: Procedure: gap filling; Procedure: connective tissue graft
- group 2: socket with damaged buccal bone plate
  Interventions: Procedure: flap elevation and guided bone regeneration; Procedure: gap filling; Procedure: connective tissue graft

INTERVENTIONS:
Procedure: flap elevation and guided bone regeneration — to rebuild the alveolar ridge convexity
  Groups: group 2
Procedure: gap filling — to use biomaterials to fill the jumping gap
Procedure: connective tissue graft — to change the soft tissue phenotype by connective tissue graft

SUMMARY:
Immediate implant placement has been advantageous in terms of reduced treatment time and fewer surgical interventions. Given the fact that the level of buccal bone acts as a major prognostic factor for IIP, the indications for immediate implant placement were suggested to be limited to intact alveolar sockets.In recent years, many attempts have been performed to compensate for the alveolar ridge resorption in immediate implant placement in compromised sockets. The clinical outcomes of IIP with guided tissue regeneration and connective tissue grafting using papilla preservation technique in compromised extraction sockets has not been previously reported.

ELIGIBILITY:
Inclusion Criteria:

* patients with anterior failing teeth (from cainine to cainine) with the presence of neighbouring teeth
* sufficient bone volume to achieve primary stability at implant insertion

Exclusion Criteria:

* with uncontrolled periodontitis
* heavy smoker (>10 cigarettes/day)
* unwilling to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in need of single implant replacement
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
mucosa recession | baseline to 1-year
  The height of the crown was measured by a peridontal probe in mid-facial aspect. The difference of the height of the crown over time was calculated as mucosa recession

SECONDARY OUTCOMES:
probing depth | baseline to 1-year
  peri-implant probing depth detected by periodontal probe examined by a peridontal probe at six sites around the crown
bleeding on probing | baseline to 1-year
  percentage of sites with bleeding on probing examined by a peridontal probe at six sites around the crown
Pink Esthetic Score (0-14) | baseline to 1-year
  Seven parameters were assessed:mesial papilla, distal papilla, soft tissue level, soft tissue contour, alveolar process deficiency, soft tissue color, and soft tissue texture. Each parameter was scored as 2,1,0.
thickness of buccal bone plate | baseline to 1-year
  the distance between the implant's facial contour and the outside surface of the buccal bone measured by cone beam computor tomograph.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hositpal, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided